CLINICAL TRIAL: NCT04258371
Title: DAPAgliflozin Sodium Water glucosE EffecTs in Patients at High Cardiovascular Risk
Acronym: DAPA-SWEET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); MOUNT SINAI HOSPITAL (Other)
Responsible Party: Principal Investigator, David Z.I. Cherney, Associate Professor of Medicine, Clinician Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-5597
Record Dates: First submitted 2020-01-23; First posted 2020-02-06 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Risk Factor
Keywords: SGLT2 inhibition; Cardiovascular risk; Dapagliflozin
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to 10mg PO dapagliflozin daily or matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin Treatment Arm (Experimental): Dapagliflozin Tablets Total Dose 10mg daily for 12 weeks
  Interventions: Drug: Dapagliflozin 10 MG
- Placebo Arm (Placebo Comparator): Placebo Matching Dapagliflozin Tablet for 12 weeks
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Dapagliflozin 10 MG — Dapagliflozin Tablets Total Dose 10mg daily for 12 weeks
  Arms: Dapagliflozin Treatment Arm
Drug: Placebo oral tablet — Placebo once daily for 12 weeks
  Arms: Placebo Arm

SUMMARY:
This study aims to elucidate the impact of SGLT2 inhibition on peripheral vascular function, renal function, fluid volume, neurohormonal activation and inflammatory/fibrotic pathways in patients with T2D at high cardiovascular risk and non-T2D patients.

DETAILED DESCRIPTION:
In light of EMPA-REG OUTCOME, CANVAS Program and DECLARE trials, we aim to elucidate the impact of SGLT2 inhibition on peripheral vascular function while also exploring the effects of this therapy on renal function, fluid volume, neurohormonal activation and inflammatory/fibrotic pathways in patients with T2D at high cardiovascular risk to best replicate the patient populations in recent cardiovascular outcome trials (CVOT), who are also participating in ongoing CVOTs such as VERTIS (ertugliflozin), as well as non-T2D patients in other ongoing trials examining cardiorenal effects of these therapies. We will test the hypothesis that in a high- risk population, regardless of T2D status, SGLT2 inhibition will improve markers of arterial stiffness (decreases in pulse wave velocity and augmentation index) in the study cohort - a surrogate marker of cardiovascular risk independent of glucose lowering. In addition, dapagliflozin will improve endothelial function ("flow-mediated vasodilatation" - FMD) and increase natriuresis (fractional excretion of sodium or FENa+), thereby reducing blood pressure, without inducing renal vasoconstriction or activation of the sympathetic nervous system (SNS). Based on extensive experimental literature, we also hypothesize that SGLT2 inhibition will suppress levels of pro-inflammatory/fibrotic mediators (see below) that have been linked with progression of cardiovascular and renal disease. The systematic understanding of the effects of SGLT2 inhibitors in the setting of patients at high cardiovascular risk will enable the design of rational physiology-based strategies to decrease the burden of cardiorenal disease, which could have important clinical and research implications. Data from DAPA-SWEET will also be valuable to better understand the results of trials that include patients using SGLT2 inhibitors as primary prevention strategies, such as in DECLARE TIMI-58.

ELIGIBILITY:
Inclusion Criteria:

1. eGFR ≥30 ml/min/1.73m2
2. In patients with type 2 diabetes, HbA1c <12.0%
3. Body Mass Index (BMI) 18.5-45.0 kg/m2
4. Blood pressure < or = 160/100 at screening (sitting)
5. Stable dose of maximally tolerated ACE inhibitor, angiotensin receptor blocker or renin inhibitor for at least 30 days
6. Stable diuretic dose for at least 14 days prior to baseline study Visit
7. High cardiovascular risk: an age of 50 years or more with at least one cardiovascular coexisting condition (coronary heart disease, cerebrovascular disease, peripheral vascular disease, chronic kidney disease of stage 3 or greater, or chronic heart failure of New York Heart Association class II or III) OR an age of 60 years or more with at least one cardiovascular risk factor, as determined by the investigator (microalbuminuria or proteinuria, hypertension and left ventricular hypertrophy, left ventricular systolic or diastolic dysfunction, or an ankle-brachial index [the ratio of the systolic blood pressure at the ankle to the systolic blood pressure in the arm] of less than 0.9).

Exclusion Criteria:

1. Type 1 Diabetes
2. Iodine intolerance
3. Hypersensitivity or allergy to dapagliflozin
4. Use of an SGLT2 inhibitor within 30 days
5. Leukocyte and/or nitrite positive urinalysis that is untreated
6. Severe hypoglycaemia within 1 month prior to screening
7. Unstable coronary artery disease with acute coronary syndrome, percutaneous intervention or bypass surgery within 3 months
8. Clinically significant valvular disease in the opinion of the investigator
9. Congestive heart failure secondary to an infiltrative cardiomyopathic process (for example amyloid) or pericardial constriction
10. Bariatric surgery or other surgeries that induce chronic malabsorption within 1 year;
11. Anti-obesity drugs or diet regimen and unstable body weight three months prior to screening;
12. Treatment with systemic corticosteroids
13. Blood dyscrasias or any disorders causing hemolysis or unstable red blood cells
14. Pre-menopausal women who are nursing, pregnant, or of child-bearing potential and not practicing an acceptable method of birth control
15. Participation in another trial with an investigational drug within 30 days of informed consent
16. Alcohol or drug abuse within three months prior to informed consent that would interfere with trial participation or any ongoing clinical condition that would jeopardize subject safety or study compliance based on investigator judgement
17. Liver disease, defined by serum levels of alanine transaminase, aspartate transaminase, or alkaline phosphatase >3 x upper limit of normal as determined during screening
18. Medical history of cancer or treatment for cancer in the last five years prior to screening, aside from uncomplicated basal cell or squamous cell carcinoma;
19. Unstable or rapidly progressive renal disease as per investigator judgement
20. Intolerance or sensitivity to SGLT2 inhibitors

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness | Acute (1 week)
  Measured using a Sphygmocor device
Arterial stiffness | Chronic (12 weeks)
  Measured using a Sphygmocor device

SECONDARY OUTCOMES:
Glomerular filtration rate | Glomerular Filtration Rate (GFR, based on plasma iohexol clearance) will be measured at 2 time points: acute (1 week) and chronic (12 weeks)
  GFR
Flow mediated dilation | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  FMD
Nitroglycerin mediated dilation | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
Systolic blood pressure | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
Diastolic blood pressure | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
Heart rate | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
Echocardiography | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Changes to systolic and diastolic function
Non-Invasive Cardiac Output Monitoring (Measured using a NICOM device) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Cardiac output and systemic vascular resistance
Bioimpedence spectroscopy | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Measure of extracellular water
Plasma concentration of natriuretic peptides | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
Plasma concentration of the renin-angiotensin aldosterone system (RAAS) hormones | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
Nitric oxide | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
Fractional excretion of sodium, using lithium clearance as a surrogate for proximal tubular sodium handling | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
Urinary concentration of the renin-angiotensin aldosterone system (RAAS) markers | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
Urinary adenosine | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
mRNA expression of monocyte chemoattractant protein-1(MCP-1) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Measured in urine and skin biopsy samples
mRNA expression of intercellular adhesion molecule-1(ICAM-1) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Measured in urine and skin biopsy samples
mRNA expression of plasminogen activator inhibitor-1(PAI-1) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Measured in urine and skin biopsy samples
mRNA expression of transforming growth factor-beta (TGF-beta) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Measured in urine and skin biopsy samples
mRNA expression of connective tissue growth factor (CTGF) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Measured in urine and skin biopsy samples
mRNA expression of interleukins (IL-1beta, IL-6) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Measured in urine and skin biopsy samples
mRNA expression of tumour necrosis factor-alpha (TNF-alpha) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Measured in urine and skin biopsy samples
mRNA expression of matrix metalloproteinases 2 (MMP2) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Measured in urine and skin biopsy samples
mRNA expression of matrix metalloproteinases 9 (MMP9) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Measured in urine and skin biopsy samples
mRNA expression of advances glycation end-product (AGE) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Measured in urine and skin biopsy samples
mRNA expression of receptor for AGE (RAGE) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
  Measured in urine and skin biopsy samples
Urinary thiobarbituric acid reactive substances (TBARS) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)
Urinary 8-hydroxydeoxyguanosine (8-OHdG) | Outcome will remeasured at 2 time points: acute (1 week) and chronic (12 weeks)

OTHER OUTCOMES:
Number of hypoglycaemic episodes | Throughout study completion, an average of 12 weeks
Serious adverse events | Throughout study completion, an average of 12 weeks
Drug related adverse events | Throughout study completion, an average of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David ZI Cherney, MD PhD FRCPC, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- Renal Physiology Laboratory, Toronto, Canada

REFERENCES:
- [Derived] Sridhar VS, Kugathasan L, Lytvyn Y, Deng Y, Liu H, Lovblom LE, Tse J, Nardone M, Floras JS, Osuntokun T, Tobushi T, Lam RCY, Lam B, Stevens J, Burger D, Touw DJ, Heerspink HJL, Lovshin JA, Perkins BA, Cherney DZI. Cardiovascular-Kidney Effects of Dapagliflozin in Patients at Cardiovascular Risk With or Without Type 2 Diabetes: Results of a Randomized, Double-Blind, Placebo-Controlled Trial. Hypertension. 2026 Feb;83(2):e25955. doi: 10.1161/HYPERTENSIONAHA.125.25955. Epub 2025 Dec 5. PMID 41347301